CLINICAL TRIAL: NCT02490163
Title: Comparison of Two Automated Mononuclear Collection Systems (Spectra Optia CMNC and MNC) in Patients Undergoing Extracorporeal Photochemotherapy. A Cross-over Equivalence Study.
Brief Title: Comparison of Two Automated Mononuclear Collection Systems in Patients Undergoing Extracorporeal Photochemotherapy. A Cross-over Equivalence Study. (MNC_CMNC)
Acronym: CMNC_MNC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Claudia Del Fante, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: doc20150414113301_CDF
Record Dates: First submitted 2015-05-28; First posted 2015-07-03 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: GvHD; Lung Graft Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CMNC (Experimental): the very recently released Spectra Optia CMNC (developed especially to collect stem cells that reside in the MNCs layer) is able to collect MNCs by continuous flow.
  Interventions: Device: Spectra Optia
- MNC (Active Comparator): The Spectra Optia MNC collects MNCs by intermittent flow: MNCs accumulate and are flushed from a secondary chamber at intervals during the procedure.
  Interventions: Device: Spectra Optia

INTERVENTIONS:
Device: Spectra Optia — The Spectra Optia® Apheresis System is an automated centrifugal system that separates whole blood into its cellular and plasma components. The device is comprised of three major sub-systems, 1) the apheresis machine itself, 2) a sterile, single-use, disposable blood tubing set, and 3) embedded software.
  Terumo BCT developed a completely automated apheresis system: the Spectra Optia MNC and CMNC based on an automatic interface-controlled technology that allows MNCs collection without the intervention of an operator. The optical sensors continuously control and adjust the buffy coat layer by adjusting the plasma flow.
  The Spectra Optia MNC collects MNCs by intermittent flow: MNCs accumulate and are flushed from a secondary chamber at intervals during the procedure. On the other hand, the very recently released Spectra Optia CMNC (developed especially to collect stem cells that reside in the MNCs layer) is able to collect MNCs by continuous flow.
  Other Names: Terumo BCT

SUMMARY:
In a study performed in 2012, the investigators demonstrated that in ECP setting , the new automated device (Spectra Optia-MNC) released by Terumo BCT for MNCs collection based on intermittent flow is safe and ensures high-quality MNC collection and yield.(5, 6) More recently (in 2013), Terumo BCT released another automated system that allows to collect stem cells and MNCs basing on a continuous collection flow.(7, 8) The aim of this cross-over study is to compare yield (i.e. collection efficiency, CE) and quality (i.e. purity and contamination) of MNCs collected from patients undergoing ECP with two different automated systems: MNC and CMNC (Terumo BCT) processing 1.5 blood volumes during every collection procedure.

DETAILED DESCRIPTION:
Two-sequences-in-four-periods cross-over, with the same patients randomized to both devices within each ECP cycle in two consecutive cycles, open-label.

Cycle 1 Cycle 1 Cycle 2 Cycle 2 Day 1 Day 2 Day 1 Day 2 Sequence A CMNC MNC MNC CMNC Sequence B MNC CMNC CMNC MNC There might be some carry over effect between procedure 1 and 2 within each cycle, because during the procedure the patient is administered fluids, and therefore cell counts/ml in the second day might be lower than in the first day; this it is intrinsic to the clinical procedure and can not be modified, but will be taken into account in statistical analyses. Carry over effect between first and second cycle is not expected, since they are performed at least 7 days apart; this allow the patient's cell blood count to be restored to baseline values; however, this will also be considered in statistical analyses.

ELIGIBILITY:
adult (>18 years) patients undergoing extracorporeal photochemotherapy for either CLAD or GvHD Inclusion criteria: age >18 years on extracorporeal photochemotherapy for either CLAD or GvHD exclusion criteria: age <18 years,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Yield of MNCs | on average at 1 month from ECP start
  absolute number of MNC/ml in bag

SECONDARY OUTCOMES:
Collection efficiency (%) | on average at 1 month from ECP start
  MNC Collection efficiency %
purity | on average at 1 month from ECP start
  percentage of MNC/ml in bag content
safety as change in platelet count in peripheral blood | single timepoint point: 10 minutes after MNC collection
  patient's platelet loss

OTHER OUTCOMES:
Yield of MNCs in GvDH vs CLAD | on average at 1 month from ECP start
  absolute number of MNC/ml in bag in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinic San Matteo Foundation, Pavia, Italy